CLINICAL TRIAL: NCT06133166
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of EG017 Ointment for the Treatment of Dry Eye in Postmenopausal Women
Brief Title: A Study for the Treatment of Dry Eye in Postmenopausal Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GenSci100-202
Record Dates: First submitted 2023-11-03; First posted 2023-11-15 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-06

CONDITIONS: Postmenopausal Women With DED

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- EG017 ointment 3% (Experimental): 60 subjects，Apply once a night on the skin side of both eyelids at bedtime, approximately 100 mg/eye per dose, for 8 weeks
  Interventions: Drug: EG017 ointment
- EG017 ointment 5% (Experimental): 60 subjects，Apply once a night on the skin side of both eyelids at bedtime, approximately 100 mg/eye per dose, for 8 weeks
  Interventions: Drug: EG017 ointment
- EG017 ointment 9% (Experimental): 60 subjects，Apply once a night on the skin side of both eyelids at bedtime, approximately 100 mg/eye per dose, for 8 weeks
  Interventions: Drug: EG017 ointment
- Placebo A (Placebo Comparator): 40 subjects，Apply once a night on the skin side of both eyelids at bedtime, approximately 100 mg/eye per dose, for 8 weeks
  Interventions: Drug: EG017 ointment placebo
- Placebo B (Placebo Comparator): 20 subjects，Apply once a night on the skin side of both eyelids at bedtime, approximately 100 mg/eye per dose, for 8 weeks
  Interventions: Drug: EG017 ointment placebo

INTERVENTIONS:
Drug: EG017 ointment — Apply once a night on the skin side of both eyelids at bedtime, approximately 100 mg/eye per dose, for 8 weeks
  Arms: EG017 ointment 3%; EG017 ointment 5%; EG017 ointment 9%
Drug: EG017 ointment placebo — Apply once a night on the skin side of both eyelids at bedtime, approximately 100 mg/eye per dose, for 8 weeks
  Arms: Placebo A; Placebo B

SUMMARY:
A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of EG017 Ointment for the Treatment of Dry Eye in Postmenopausal Women

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of EG017 ointment for the treatment of DED in postmenopausal women

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old；
2. Postmenopausal women
3. Diagnosed with DED for at least 6 months;
4. If receiving artificial tears for DED, discontinue use 1 day prior to baseline exam; if receiving other topical medications for DED, discontinue use more than 1 week or 5 half-lives (whichever is longer) prior to baseline exam; willing to discontinue use of any other topical medication for DED other than artificial tears for the entire study period;

6） Voluntarily participate in the trial, understand and sign written informed consent, and be willing and able to comply with the clinical trial arrangements

Exclusion Criteria:

1. Presence of a history of allergic reactions to the study drug, similar drugs or ingredients;
2. DED secondary to scar formation (e.g., radiation therapy, alkali burns, Stevens-Johnson syndrome, scar-like aspergillosis) or conjunctival cupped cell destruction (e.g., vitamin A deficiency);
3. Screening slit lamp examinations reveal clinically significant ocular disease or abnormalities in the ocular anatomy
4. Schirmer test (without anesthesia) < 3mm/5min；
5. Screening stage CFS revealed a lamellar defect in the corneal epithelium or ≥ 2 areas of corneal staining fusion > 50%;
6. BCVA ≤ 0.2 in both eyes during the screening period;
7. Presence of active ocular or periocular acne, ocular allergies and ocular infections at the time of screening, which in the judgment of the investigator may interfere with the test;
8. History of corneal contact lens wear within 1 month prior to screening, or inability to stop wearing corneal contact lenses during the screening period to the end of the study;
9. History of treatment with topical steroids, topical NSAIDs, topical cyclosporine, lifitegrast, tacrolimus, serum tears, or topical antiglaucoma medications within 1 month prior to screening;
10. Have received or had removed a permanent lacrimal embolus within 1 month prior to screening, or plan to have a lacrimal embolus installed or related to removal of a lacrimal embolus during the study, or plan to have a lacrimal embolus lysed during the study;
11. LipiFlow treatment within 3 months prior to screening, or intense pulsed light treatment within 1 month prior to screening, or blepharoplasty within 1 week prior to screening;
12. History of intraocular surgery or ocular laser surgery within 6 months prior to screening, or planned ocular or eyelid surgery during the study period;
13. Presence of a history of herpetic keratitis, ocular or periocular malignancy;
14. Presence of an infection requiring systemic antibiotic (including antibacterial, antiviral, antifungal) control within 7 days prior to screening;
15. Severe systemic autoimmune diseases;
16. Presence of the clinically significant diseases；
17. Participated in other drug or device clinical trials within 1 month prior to screening;
18. Any medical or other condition that the investigator believes may affect the clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-09 (Estimated)

PRIMARY OUTCOMES:
tCFS | 8 weeks
  Change from baseline in tCFS（Total corneal fluorescein staining）after 8-week of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Xiamen Ophthalmology Center Affiliated to Xiamen University, Xiamen, Fujian, China